CLINICAL TRIAL: NCT06834737
Title: Understanding Endometriosis-related Symptoms and Their Relationship to Sleep
Brief Title: The Sleep-pain Relationship in Women with Endometriosis
Acronym: ENDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Olivier Mairesse, Professor, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2526_ENDO
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: ESM; Endometriosis; Sleep; Cyclic pain; Chronic pelvic pain
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclic pain (Other): Women eligible for the study are adult, non-(post)menopausal individuals who have received a laparoscopic and histopathological diagnosis of en-dometriosis. They have been experiencing cyclic pain (before, during, and/or after menstruation or monthly flare-ups without menstruation) for at least two months. Participants do not expect to undergo gynecologic or other surgical procedures for en-dometriosis during the study period and are not pregnant or breastfeeding. They must have no external factors interfering with their sleep for three or more nights per week, such as work, noise, or caregiving responsibilities.
  intervention: 6 item diary twice a day over the course of 2 months.
  Interventions: Other: ecological sampling method
- Non-cyclical pain (Other): Women eligible for the study are adult, non-(post)menopausal individuals who have received a laparoscopic and histopathological diagnosis of en-dometriosis. They have been experiencing non-cyclic pain for at least six months. Participants do not expect to undergo gynecologic or other surgical procedures for en-dometriosis during the study period and are not pregnant or breastfeeding. They must have no external factors interfering with their sleep for three or more nights per week, such as work, noise, or caregiving responsibilities.
  intervention: 6 item diary twice a day over the course of 2 months.
  Interventions: Other: ecological sampling method

INTERVENTIONS:
Other: ecological sampling method — 6-item diary, twice a day, over the course of 2 months.

SUMMARY:
The goal of this study is to examine the sleep-pain relationship in women diagnosed with endometriosis, by monitoring different symptoms of endometriosis and sleep through an experience sample method study (ESM).The main question it aims to answer is:

How does sleep impact cyclic and chronic pain and vice versa in women with endometriosis?

Participants will be asked to fill in a 6-item diary (twice a day) over the course of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult premenopausal women with a laparoscopic and histopathological diagnosis of endometriosis, without a history of hysterectomy, experiencing cyclic or chronic pelvic pain for 3 months or longer, with pain intensity of at least 3 out of 10 over the past 3 months, experiencing non-restorative sleep (defined as a subjective feeling of being unrefreshed up-on awakening) for 3 months or longer, in the absence of elevated risk for intrinsic sleep disorders (such as sleep apnea or restless leg syndrome), and having sufficient knowledge of either French, Dutch, or English

Exclusion Criteria:

* Participants younger than 18 years old, without laparoscopic and histopathological diagnosis of endometriosis, participants with a hysterectomy or pain intensity lower than 3/10, with restorative sleep or sleep apnea and restless leg syndrome, shift work and insufficient knowledge of either French, Dutch or English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | From enrollment to the end of ESM at 8 weeks
  Morning assessment: Irrespective of how much you slept, how good was the quality of your sleep? (0= not at all, 7= very good).
Pain intensity | From enrollment to the end of ESM at 8 weeks
  Evening assessment: How much pain did you experience today? (0= none, 7= very much)

SECONDARY OUTCOMES:
Mood | From enrollment to the end of ESM at 8 weeks
  Evening assessment:
  How good was your mood overall today? (0= No good mood at all, 7= very good)
Stress | From enrollment to the end of ESM at 8 weeks
  Evening assessment:
  How much stress did you experience today? (0= none, 7= very much)
Sleep duration + sleep regulariy | From enrollment to the end of ESM at 8 weeks
  Morning assessment:
  1. What time did you go to bed last night?
  2. What time did you wake up this morning?
  3. For how long were you awake during the night?
  Sleep duration will be calculated based on Q1,Q2,Q3. Sleep regularity will be calculated based on Q1, Q2.
Fatigue | From enrollment to the end of ESM at 8 weeks
  Evening assessment:
  How fatigued were you today? (0= Not at all, 7= very fatigued)
Cognitive performance | From enrollment to the end of ESM at 8 weeks
  Evening assessment:
  How well do you think you performed cognitively today? (0= Not at all, 7= very good)
Night pain | From enrollment to the end of ESM at 8 weeks
  Morning assessment: How much pain did you experience last night? (0= none, 7= very much)
Pain frequency | From enrollment to the end of ESM at 8 weeks
  Evening assessment: How often did you experience pain today? (0 = not at all, 7 = continuous)

OTHER OUTCOMES:
Menstrual cycle | From enrollment to the end of ESM at 8 weeks
  Evening assessment: Have you menstruated today or experienced menstrual-like symptoms (e.g., spotting/intermittent bleeding,...)?
  * Yes
  * No
  * Not applicable
Morning/ evening pain | From enrollment to the end of ESM at 8 weeks
  Morning and evening assessment:
  How much pain do you experience right now? (0= none, 7= very much)
Medication intake | From enrollment to the end of ESM at 8 weeks
  Did you take any medication or other substances today? If so, please specify the medication and dosage (example: '1g dafalgan')
  * No
  * Yes, sleep medication ______
  * Yes, pain medication _______
  * Yes, sedatives ________
  * Yes, other ________

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunes FR, Ferreira JM, Bahamondes L. Pain threshold and sleep quality in women with endometriosis. Eur J Pain. 2015 Jan;19(1):15-20. doi: 10.1002/ejp.514. Epub 2014 Apr 14. PMID 24733758
- [Background] Arion K, Orr NL, Noga H, Allaire C, Williams C, Bedaiwy MA, Yong PJ. A Quantitative Analysis of Sleep Quality in Women with Endometriosis. J Womens Health (Larchmt). 2020 Sep;29(9):1209-1215. doi: 10.1089/jwh.2019.8008. Epub 2020 Mar 13. PMID 32176592
- [Background] Chaichian S, Mehdizadehkashi A, Haghgoo A, Ajdary M, Derakhshan R, Rokhgireh S, Sarhadi S, Nikfar B. Sleep disorders in patients with endometriosis; a cross-sectional study. BMC Womens Health. 2024 Jun 14;24(1):340. doi: 10.1186/s12905-024-03185-x. PMID 38877485
- [Background] Sumbodo CD, Tyson K, Mooney S, Lamont J, McMahon M, Holdsworth-Carson SJ. The relationship between sleep disturbances and endometriosis: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2024 Feb;293:1-8. doi: 10.1016/j.ejogrb.2023.12.010. Epub 2023 Dec 9. PMID 38091847